CLINICAL TRIAL: NCT00001216
Title: Non-Invasive Stimulation of the Human Central Nervous System (Digitimer)
Brief Title: Non-Invasive Electrical Stimulation of the Human Brain
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 860020; 86-N-0020
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-12

CONDITIONS: Cerebrovascular Disorders; Healthy; Nervous System Diseases; Spinal Cord Injuries
Keywords: Amputations; Brainstem Stimulation; Cerebellar Stimulation; Cortical Motor Physiology; Electrical Stimulation; Motor Cortex; Plasticity; Spinal Cord Injury; Stroke
MeSH Terms: conditions — Cerebrovascular Disorders; Nervous System Diseases; Spinal Cord Injuries; Stroke

SUMMARY:
This study is designed to allow researchers to use transelectrical stimulation to explore the function of the human nervous system and improve diagnosis of neurological disorders.

Transcranial electrical stimulation is a non-invasive technique that can be used to stimulate brain activity and gather information about brain function. Electrical stimulation involves placing electrodes on the scalp or skin and passing an electrical current between them. When this is done, an electrical field is created that activates areas of the brain that control muscles. Muscle activity as a result of the stimulation can be recorded and analyzed.

DETAILED DESCRIPTION:
This protocol application is written to permit us to use transcranial electrical stimulation, a safe and noninvasive method for activating the brain, spinal cord, or proximal nerves through the skin, in appropriate subjects. We will use this technique to explore the function of the human central and peripheral nervous system and to aid in the diagnosis of neurological disorders.

ELIGIBILITY:
Males and females, ages 18 and over.

Diverse racial groups.

Amputees and others with whom we will have no patient-care relationship may also be considered to be volunteers.

Patients will be recruited from those referred to the Human Motor Control Section, NINDS who have neurological syndromes that are of interest.

On rare occasions we may attempt to study children as young as 10 years with TES.

Individuals without indwelling cardiac lines and pacemakers.

Patients recruited for study would come from those referred to the EMG laboratory and to the Human Motor Control Clinic who would have distinct neurologic syndromes from well defined peripheral and central nervous system lesions including hemiplegia from stroke, trauma, tumor or focal demyelination (most commonly patients would have hemiplegia from stroke), peripheral nerve lesions, amputations, spinal cord injury.

Normal volunteers, including NIH employees, would be healthy adults without history of physical examination evidence of neurologic disease and individuals with different types of amputations involving upper and lower extremities.

Volunteers may also be participants in the electrophysiological protocol (84-N-0196).

No history of epilepsy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 175
Dates: Start 1986-02; Study Completion 2001-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Cohen LG, Meer J, Tarkka I, Bierner S, Leiderman DB, Dubinsky RM, Sanes JN, Jabbari B, Branscum B, Hallett M. Congenital mirror movements. Abnormal organization of motor pathways in two patients. Brain. 1991 Feb;114 ( Pt 1B):381-403. doi: 10.1093/brain/114.1.381. PMID 2004248
- [Background] Brasil-Neto JP, Pascual-Leone A, Valls-Sole J, Cammarota A, Cohen LG, Hallett M. Postexercise depression of motor evoked potentials: a measure of central nervous system fatigue. Exp Brain Res. 1993;93(1):181-4. doi: 10.1007/BF00227794. PMID 8467889
- [Background] Brasil-Neto JP, Cohen LG, Pascual-Leone A, Jabir FK, Wall RT, Hallett M. Rapid reversible modulation of human motor outputs after transient deafferentation of the forearm: a study with transcranial magnetic stimulation. Neurology. 1992 Jul;42(7):1302-6. doi: 10.1212/wnl.42.7.1302. PMID 1620338